CLINICAL TRIAL: NCT00093288
Title: A Multi-Centre, Randomised, Double-Blind, Parallel-Group, Placebo-Controlled, Flexible Dose Study to Evaluate the Efficacy, Safety and Tolerability of Extended-release Bupropion Hydrochloride (150mg-300mg Once Daily) in Elderly Subjects With Major Depressive Disorder
Brief Title: Major Depressive Disorder In The Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK130940
Record Dates: First submitted 2004-10-05; First posted 2004-10-07 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Depressive Disorder, Major
Keywords: MDD; bupropion; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

INTERVENTIONS:
Drug: bupropion XL

SUMMARY:
This is a placebo-controlled study evaluating the effectiveness of medication in elderly subjects with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Major Depressive Disorder with DSM-IV criteria for their current episode for at least 8 weeks.

Exclusion Criteria:

* Patient has current or past history of seizure disorder or brain injury.
* Patient has a diagnosis of anorexia or bulimia within the past 12 months.
* Patient has a past or current DMS-IV diagnosis of schizophrenia or any other psychotic disorder(s).
* Patient has had a myocardial infarction within 1 year or a history of uncontrolled hypertension or unstable heart disease with 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 364
Dates: Start 2004-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale Clinical Global Impression Improvement Scale Clinical Global Impression Severity Scale Hamilton Anxiety Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Australia (4):
  - GSK Investigational Site, Caboolture, Queensland
  - GSK Investigational Site, Everton Park, Queensland
  - GSK Investigational Site, New Farm, Queensland
  - GSK Investigational Site, St Albans, Victoria
- Belgium (3):
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Mont-Godinne
  - GSK Investigational Site, Montignies-sur-Sambre
- GSK Investigational Site, Mikkeli, Finland
- Netherlands (5):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Grubbenvorst
  - GSK Investigational Site, Hilversum
  - GSK Investigational Site, Hoogvliet
  - GSK Investigational Site, Wildervank
- GSK Investigational Site, Oslo, Norway
- GSK Investigational Site, Moscow, Russia